CLINICAL TRIAL: NCT04847154
Title: Endometrium Microbiome Alterations in Cesarean Section Diverticula Before and After Transvaginal Repair Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-003
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study compares the microbiome differences in the endometrium between normal people and patients with uterine diverticula after cesarean section and aims to discover the essential microbes and their metabolites that highly associate with the repair of myometrium through metagenomics and metabolomics. It verifies that flora disorder in the endometrium is the important cause of poor uterine repair after cesarean section. Then these patients with uterine diverticula receive the transvaginal repair surgery. Through the follow-up with them, we gain the microbiome differences of the endometrium before and after the surgery and show the validity of transvaginal repair surgery in the level of microbiome and metabolism.

ELIGIBILITY:
Inclusion Criteria:

have one cesarean delivery, have intermenstrual spotting after the cesarean section or Residual muscle thickness was less than 3.0 mm at the preoperative stage underwent magnetic resonance imaging and transvaginalultrasound to evaluate the size of the defect and the Residual muscle thickness before surgery have vaginal repair of Cesarean Section Diverticula write consent for operation.

Exclusion Criteria:

have a history of endocrine disorders have coagulation disorders use of intrauterine devices have sub-mucous myoma have endometrial diseases have endometrial cysts, uterine fibroids, and adenomyosis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 Healthy women with cesarean section without Cesarean Section Diverticula 30 Healthy women with cesarean section with Cesarean Section Diverticula
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-12 (Estimated); Primary Completion 2021-04-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Endometrium Microbiome | In the 7th day of the period
  analysis the microbiome differences in the endometrium between normal people and patients with uterine diverticula after cesarean section and after vaginal repair surgery